



## Human Milk Lipid Profile Assessment and Influences of Mother's Diet

## INFORMED CONSENT

This form must be signed by you only if you decide to participate in the study. You can withdraw your consent at any time.

I declare to receive a signed copy of this consent form together with a dated and signed copy of the information sheet. I also declare:

- to have received from the investigator exhaustive explanations regarding the request for participation in the study, in particular on the purposes and procedures;
- having read and understood the information sheet that was given to me sufficiently in advance and confirming what was explained to me;
- having had the opportunity to ask questions and have received satisfactory answers;
- take charge of the delivery of the letter relating to the study to my attending physician;
- be aware that participation is voluntary, with the assurance that the refusal to participate will in no way affect the quality of the assistance received;
- be aware that, if I withdraw my consent, the data collected before the withdrawal of consent will be used by the researchers;
- to consent and authorize the collection and processing of my personal data, pursuant to Legislative Decree n. 196/2003 (privacy code), for the purposes of the research within the limits and with the methods indicated in the information provided with this document.